CLINICAL TRIAL: NCT02436603
Title: Integrative Approaches to Managing Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 010-15
Record Dates: First submitted 2015-04-28; First posted 2015-05-07 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Irritable Bowel Syndrome; IBS
Keywords: Irritable Bowel Syndrome; IBS; Mind-Body Training; Integrative Medicine; FODMAP
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutrition/Mind-Body Coaching (Other): The intervention will consist of weekly group sessions lasting 75-90 minutes during which participants will receive training in the FODMAP diet and mind-body skills.
  Interventions: Behavioral: Nutrition/Mind-Body Coaching
- Waitlist Control Group (No Intervention): Waitlist subjects. At the end of the 12-week study period, waitlist subjects will be offered the four-week nutrition and mind-body intervention.

INTERVENTIONS:
Behavioral: Nutrition/Mind-Body Coaching — Following the four-week treatment intervention, participants will then be enrolled in an 8-week health coaching follow-up period. During this time participants will have a 45-60 minute telephone session with a health coach weekly for two weeks, then biweekly for four weeks.
  Arms: Nutrition/Mind-Body Coaching

SUMMARY:
The purpose of this project is to examine whether a low cost, group-oriented integrative medicine approach to irritable bowel syndrome improves participant outcomes. The intervention will combine nutrition counseling on the low FODMAP diet (decreased grains and other disaccharides) and mind-body training with follow-up health coaching.

These participants will be randomized to either a 4-week group-oriented treatment intervention incorporating a low FODMAP (fermentable oligosaccharides, disaccharides, monosaccharides and polyols) diet and mind-body therapies followed by an 8-week health coaching follow-up period or a waitlist control group. At the end of the 12-week study period, waitlist subjects will be offered the four-week nutrition and mind-body intervention. Over the 12-week study period, we will examine and report on the impact of this treatment intervention on IBS symptoms and quality of life in this population. The investigators will collect data on IBS outcomes as well as on depression and stress.

DETAILED DESCRIPTION:
This project will test the effectiveness of an integrative medicine approach in treating irritable bowel syndrome (IBS). Over the course of 18 months, we will recruit 85 participants with IBS in New York City. These participants will be randomized to either a 4-week group-oriented treatment intervention incorporating a low FODMAP (fermentable oligosaccharides, disaccharides, monosaccharides and polyols) diet and mind-body therapies followed by an 8-week health coaching follow-up period or a waitlist control group. At the end of the 12-week study period, waitlist subjects will be offered the four-week nutrition and mind-body intervention. Over the 12-week study period, we will examine and report on the impact of this treatment intervention on IBS symptoms and quality of life in this population. The investigators will collect data on IBS outcomes as well as on depression and stress.

The hypothesis is that participants will report decreased symptoms and improved function and quality of life as a result of the four-week nutrition and mind-body intervention and 8-week health coaching follow-up period. The goal of this project is to develop a low-cost, effective integrative intervention for IBS, which can be replicated in settings across the U.S.

Objectives The purpose of this project is to examine whether a low cost, group-oriented integrative medicine approach to irritable bowel syndrome improves participant outcomes. The intervention will combine nutrition counseling on the low FODMAP diet and mind-body training with follow-up health coaching.

The hypothesis is that participants will report decreased symptoms as measured by the IBS Symptom Severity Score and improved function and quality of life as a result of the intervention when compared to usual care.

Background Irritable bowel syndrome (IBS) is a chronic debilitating functional gastrointestinal disorder that has a profound effect on the quality of life (QOL) of individuals with IBS. The estimated prevalence of IBS in the general population ranges from 3% to 20%, with most studies estimating that IBS affects 10% to 15% of the general population. Despite its high level of prevalence, the exact causes of IBS are not well understood. Researchers believe that IBS is caused by a wide variety of mental and physical health problems including hypersensitivity, brain-gut signal issues, bacterial gastroenteritis, depression, anxiety, food sensitivity, body chemical imbalances, and/or genetics.

Background: Low FODMAP Diet for IBS More than 60% of IBS patients report worsening of symptoms after meals, 28% of these within 15 minutes after eating and 93% within 3 hours. The role of diet in inducing or exacerbating IBS systems has been explored for decades. Numerous studies have examined the role of lactose intolerance and fructose malabsorption in IBS. Additional research on oligosaccharides and the incompletely absorbed sugar alcohol polyols, sorbitol, and mannitol, has revealed a role in IBS symptoms. Grouping of these poorly absorbed, short chain carbohydrates- fermentable oligosaccharides, disaccharides, monosaccharides and polyols- according to their chain length resulted in the acronym FODMAP, and in 2005, the first paper describing the FODMAP hypothesis was published. Evidence continues to accumulate that the consumption of FODMAPs may contribute to symptoms in individuals with IBS.

FODMAPs are poorly absorbed, osmotically active, and increase delivery of water and fermentable substrates to the proximal colon and are rapidly fermented by bacteria. The poor absorption and fermentation of the short chain carbohydrates contributes to the bloating, distension, abdominal pain, and flatulence of individuals with IBS. In a comparison of standard dietary advice versus FODMAP for individuals with IBS, a low FODMAP diet showed significantly greater reduction in abdominal pain, bloating, and flatulence compared to the standard dietary advice group. A high FODMAP diet altered the pattern of gas production, induced prolonged hydrogen production in the intestine that was greater in individuals with IBS versus healthy controls, influenced the amount of methane produced, and induced gastrointestinal and systemic symptoms in individuals with IBS. A low FODMAP diet reduced abdominal pain, bloating, flatulence, and diarrhea in individuals with inflammatory bowel disease. In a prospective study of 90 patients with IBS followed for 15 months, a low FODMAP diet significantly decreased abdominal pain, bloating, flatulence, and diarrhea, with greater improvement with greater dietary adherence.

Background: Mind-Body Therapies for IBS Psychological therapies or mind-body therapies such as hypnosis, biofeedback, and psychotherapy represent some of the most effective treatments for IBS and are especially useful for motivated patients with moderate to severe IBS.

The scientific evidence involving mind-body therapies for IBS began in 1927 when American researcher, Dr. Edmund Jacobson, conducted the first randomized trial using progressive relaxation for IBS treatment and found significant benefit. In recent years, a vast majority of research surrounding mind-body approaches for IBS has come from a research group at University Hospital in South Manchester, UK led by Dr. Peter Whorwell. In 1984, the Whorwell group developed a hypnosis procedure specifically for treating IBS called "gut directed hypnotherapy". The intervention consists of seven half-hour sessions of decreasing frequency. In addition, patients are all given self-hypnosis tapes for daily practice. A 2005 review published by the American Society of Clinical Hypnosis examined 14 studies measuring efficacy and mechanism of hypnosis for IBS treatment (12 of the 14 studies utilized an adaptation of the Whorwell group procedure). Based on the studies investigated, the review concluded "hypnosis consistently produces significant results and improves the cardinal symptoms of IBS in the majority of patients." A separate 2006 review conducted by researchers at the University of Birmingham in England, concluded that existing scientific evidence suggest that hypnosis is effective in the treatment and management of IBS (10 of the 18 studies examined indicated significant benefit).

Regarding long-term benefit, the existing scientific evidence is supportive of mind-body approaches for IBS treatment. A long-term follow-up study of IBS patients (n=204) treated with hypnosis revealed that of the 71% who initially responded to hypnosis, 81% maintained their improvement overtime while the remaining 19% reported only slight deterioration in their IBS symptoms. Also important was that patients reported to be using fewer medications to manage IBS following hypnosis treatment. In their conclusion, the study authors determined that the benefits of hypnosis seemed to last for up to 5 years after treatment. A 1989 comparative study from England determined that hypnosis for treatment of IBS in groups of up to 8 patients was as effective as individual therapy.

ELIGIBILITY:
Inclusion Criteria:

* IBS diagnosis> 12 months in duration
* Over 18 years of age
* English speaking

Exclusion Criteria:

* Active major psychiatric illness which would potentially interfere with participation in the study 2. Pregnancy 3. Active eating disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-04; Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
IBS Symptom Severity Scale | Baseline and week 12
  a validated tool which is currently the gold standard for evaluating interventions for IBS. Change in IBS Symptom Severity Scale at week 12 as compared to Baseline
IBS Quality of Life (IBS-QOL) | Baseline and Week 12
  Change in IBS-QOL at week 12 as compared to Baseline

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGIC) | Baseline and Week 12
  The PGIC is a single question 7-point categorical scale that captures a patient's experience of treatment. Change in PGIC at week 12 as compared to baseline.
Perceived Stress Scale (PSS) | Baseline and Week 12
  Change in Measure of Stress at week 12 as compared to baseline

OTHER OUTCOMES:
Center for Epidemiological Studies - Depression Scale (CES-D) | Baseline and Week 12
  Change in a well-validated, 20-item measure of depression at week 12 compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth McDonald, MS,RD,CSS, Principal Investigator — The Center for Health & HealingDepartment of Integrative MedicineMount Sinai Beth Israel
Locations (1):
- Center for Health and Healing, New York, New York, United States

REFERENCES:
- [Background] Grundmann O, Yoon SL. Irritable bowel syndrome: epidemiology, diagnosis and treatment: an update for health-care practitioners. J Gastroenterol Hepatol. 2010 Apr;25(4):691-9. doi: 10.1111/j.1440-1746.2009.06120.x. Epub 2010 Jan 13. PMID 20074154